CLINICAL TRIAL: NCT00853879
Title: An Exploratory, Randomized, Blinded, Placebo-Controlled Trial of Folic Acid and L-methylfolate in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCRC 0143
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Folic Acid; Vitamin B 6; Vitamin B 12; 5-methyltetrahydrofolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1. B6, B12, folate (Active Comparator): Triple therapy with folate. Intervention #1.
  Interventions: Dietary Supplement: Folic Acid, Vitamin B6, Vitamin B12
- Arm 2. B6, B12, L-methylfolate (Active Comparator): Triple therapy with L-methylfolate. Intervention #2
  Interventions: Dietary Supplement: B6, B12, L-methylfolate
- Arm 3. B6, B12, Placebo (Placebo Comparator): Triple therapy with placebo. Intervention #3.
  Interventions: Dietary Supplement: B6, B12, Placebo

INTERVENTIONS:
Dietary Supplement: Folic Acid, Vitamin B6, Vitamin B12 — Intervention #1. A combination of the following vitamin supplements: 2.5mg of folate, 25mg of vitamin B6 and 2mg of vitamin B12. This combination will be described as "triple therapy with folate."
  Arms: Arm 1. B6, B12, folate
Dietary Supplement: B6, B12, L-methylfolate — Intervention #2. A combination of the following vitamin supplements: 2.8mg of L-methylfolate, 25 mg of vitamin B6 and 2mg of vitamin B12.
  Arms: Arm 2. B6, B12, L-methylfolate
Dietary Supplement: B6, B12, Placebo — Intervention #3. A combination of the following vitamin supplements: 25mg of vitamin B6 and 2mg of vitamin B12 without supplementary folate or L-methylfolate. This combination will be described as "triple therapy with placebo"
  Arms: Arm 3. B6, B12, Placebo

SUMMARY:
This study is being conducted to assess the impact of folate and L-methylfolate on the progression of Parkinson's. The investigators are specifically looking for the effect of these nutritional supplements in Parkinson's patients who have an antibody that effects their body's utilization of folate. An antibody is a protein produced by the body's immune system to recognize foreign substances. Normally, people do not have an antibody that prevents folate from working properly in the brain but it appears that some people may have such an antibody. Folate is an important vitamin that takes part in many critical cell functions so an antibody that prevented it from entering the brain properly could cause or worsen certain neurological disorders like Parkinson's. The results of this preliminary study will help determine whether it is reasonable to proceed with further study of any of these supplements for the treatment of Parkinson's. Patients interested in participating will have a blood test to see if they have folate antibodies. Patients with the antibody will be eligible to further participate in the study. The investigators will measure the effects of folate and L-methylfolate on Parkinson's disease by measuring the change in your Parkinson's disease symptoms over three months of treatment. The investigators will also be looking at the blood of some individuals who do not have Parkinson's. This is called a control group and will allow us to compare how common the folate antibody is in the general population compared with the Parkinson's population.

ELIGIBILITY:
Inclusion Criteria:

* PD subjects:

  * Diagnosis of Parkinson's based upon the presence of 2 or more of the cardinal clinical features of the disease as determined by a movement disorders specialist.
  * Age > 30.
  * Able to provide informed consent.
  * All anti-Parkinson's medications will be permitted but all evaluations will be done in the medication OFF state (at least 12 hours following the last dose of medication).
* Healthy Controls *Age > 30

Exclusion Criteria:

* PD Subjects:

  * Age < 30.
  * Presence of concomitant active neurological disorders as deemed significant by the investigator.
  * History of clinically significant diabetes, vascular disease, renal, thyroid or hepatic dysfunction or of Leber's optic neuropathy as determined by the investigator.
  * History of significant medical illness as determined by the investigators.
  * The following medications will be excluded: thiazide diuretics, azathioprine, phenytoin, phenobarbital, primidone, sulfa-containing medications, cimetidine, anti-tuberculosis medications, methotrexate, chemotherapeutic agents and oral contraceptives.
  * Subjects taking vitamin supplementation in excess of one daily standard multivitamin.
  * Pregnancy (excluded not for perceived risk but because most pregnant women are taking supplemental folate).
* Healthy Controls:

  * Age < 30
  * Any known active neurological condition deemed significant by the investigator.
  * History of significant, active renal or hepatic dysfunction as determined by the investigator.
  * History of significant active medical illness as determined by the investigators.
  * The following medications will be excluded: thiazide diuretics, azathioprine, phenytoin, phenobarbital, primidone, sulfa-containing medications, cimetidine, anti-tuberculosis medications, methotrexate, chemotherapeutic agents and oral contraceptives.
  * Subjects taking vitamin supplementation in excess of one standard daily multivitamin.
  * Pregnancy (most pregnant women are taking folate).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
This study is being conducted to assess the impact of folate and L-methylfolate on the progression of Parkinson's. The primary endpoint variable will be the change in UPDRS from baseline to 3 months ("change score"). | 3 years

SECONDARY OUTCOMES:
Secondary endpoints will be Folate receptor autoantibody levels and plasma Hcy levels | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pourfar, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute For Medical Recearch, Manhasset, New York, United States